CLINICAL TRIAL: NCT03323541
Title: Utilisation du ZArzio® en Post-Autogreffe de Cellules Souches périphériques Des Patients Atteints de Lymphome ou Myélome (in French)
Brief Title: Use of Zarzio® in Post-autologous Stem Cell Transplantation Procedure
Acronym: ZAPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ZAPA
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma; Non-hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: biosimilars; filgrastim; Stem cell transplantation; lymphoma; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma | interventions — Filgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group of patients treated with Zarxio: All consecutive patients, treated for lymphoma or myeloma, which underwent autologous stem cell transplantation in the University Hospital of Brest. All these patients were treated with biosimilars of Filgrastim: Zarzio®.
  Interventions: Drug: Filgrastim Prefilled Syringe [Zarzio®]

INTERVENTIONS:
Drug: Filgrastim Prefilled Syringe [Zarzio®] — Daily subcutaneous injection of Zarxio post ASCT, from day 5 until bone marrow recovery (neutrophils >1 giga/l)
  Other Names: Filgrastim prefilled syringe [Neupogen®]

SUMMARY:
There are limited data concerning the use of biosimilars of filgrastim in autologous stem cell transplantation (ASCT). This study aimed to evaluate G-CSF efficiency and safety (based on haemograms, transfusion needs and complications) of two biosimilars (Zarzio and Ratiograstim®) compared to those of Neupogen® for our patients who underwent ASCT.

DETAILED DESCRIPTION:
Since 2008, Investigator collected data of all patients who underwent ASCT to treat lymphoma or myeloma.

All the patients signed an institutional informed consent form before the harvest of peripheric stem cells (PROMISE program). Patients received Neupogen® (Amgen-SA) between April 2008 and February 2010, and the next group of patients was treated with Ratiograstim® (Ratiopharm GmbH) until May 2012. The last group of patients received Zarzio® (Sandoz GmbH) until November 2014.

Investigator studied the impact of the Zarzio® use on biological parameters of the bone marrow recovery, transfusion needs and infectious complications. These parameters were then compared to those of the previous patients which were treated with the two other drugs.

The patients were recruited in the University Hospital of Brest. They were consecutive patients, treated by ASCT for their high risk lymphoma and myeloma but without selection.

ELIGIBILITY:
Inclusion Criteria:

* patients with DLBCL or multiple myeloma
* patients who underwent ASCT in our hospital
* patients treated by Zarzio® in post-ASCT phase to accelerate the bone marrow recovery

Exclusion Criteria:

* patients who underwent ASCT but for other diseases
* patients who underwent ASCT for the required diseases but treated with an other biosimilar of Filgrastim
* patients who did not sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated by ASCT in the case of DLBCL or Hodgkin disease or multiple myeloma
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
time to bone marrow recovery | daily evaluation, around 8 days normally
  timing in days from the day of ASCT until the day when neutrophils >1 giga/l

CONTACTS AND LOCATIONS:
Overall Officials: IANOTTO Jean-Christophe, MD, PhD, Principal Investigator — Hématologie Clinique-Institut de Cancéro-Hématologie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nicol C, Henry C, Couturier MA, Delepine P, Tripogney C, Buors C, Guillerm G, Berthou C, Tempescul A, Ianotto JC. Biosimilars of filgrastim in autologous stem cell transplantation: certain differences for myeloma patients only. Leuk Lymphoma. 2017 Sep;58(9):1-3. doi: 10.1080/10428194.2017.1285025. Epub 2017 Feb 7. No abstract available. PMID 28278727